CLINICAL TRIAL: NCT03118167
Title: Intervention Effect of Tea Polyphenols (TP) and Water-Soluble Antioxidant Of Bamboo Leaves (AOB-w) on Short- and Long-term Internal Exposure of Acrylamide in Chinese Adolescents
Brief Title: Intervention Effect of TP and AOB-w on Acrylamide Exposure in Chinese Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Yu Zhang, Associate professor, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: RCT-001-AA
Record Dates: First submitted 2016-11-24; First posted 2017-04-18 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Intervention
Keywords: Acrylamide; Tea polyphenols; Water-soluble antioxidant of bamboo leaves
MeSH Terms: interventions — Acrylamide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tea polyphenols & Acrylamide (Experimental): TP 0.05g, 0.1g, 0.2g (starches filled, up to 0.35g) capsule by mouth, Acrylamide (Potato Chips) 12.6μg/kg b.w. by mouth, for one single oral dose
  Interventions: Dietary Supplement: Tea polyphenols; Other: Acrylamide (Potato Chips)
- AOB-w & Acrylamide (Experimental): AOB-w 0.35g capsule by mouth, Acrylamide (Potato Chips) 12.6μg/kg b.w. by mouth, for one single oral dose
  Interventions: Dietary Supplement: AOB-w; Other: Acrylamide (Potato Chips)
- Placebo & Acrylamide (Active Comparator): Placebo (Starches) 0.35g capsule by mouth, Acrylamide (Potato Chips) 12.6μg/kg b.w. by mouth, for one single oral dose
  Interventions: Other: Placebo; Other: Acrylamide (Potato Chips)

INTERVENTIONS:
Dietary Supplement: Tea polyphenols — Tea polyphenols 0.05g, 0.1g, 0.2g (starches filled up to 0.35g), edible capsule
  Other Names: TP
  Arms: Tea polyphenols & Acrylamide
Dietary Supplement: AOB-w — Water-soluble antioxidant of bamboo leaves 0.35g, edible capsule
  Other Names: Water-soluble antioxidant of bamboo leaves
  Arms: AOB-w & Acrylamide
Other: Placebo — Edible starches 0.35g, edible capsule
  Arms: Placebo & Acrylamide
Other: Acrylamide (Potato Chips) — Potato Chips bought from market, corresponding to acrylamide (12.6μg/kg b.w. )

SUMMARY:
A double-blind randomized controlled trial (RCT) was conducted in current human study. This study aims to investigate the intervention effect of AOB-w on the short-term exposure and toxicokinetics of acrylamide, a dietary hazardous substance generated during heat processing, in Chinese adolescents.

DETAILED DESCRIPTION:
In the morning of test day, participants were served with a meal of potato chips, corresponding to a single oral dose of 12.6 μg/kg b.w. exposure to acrylamide, and an edible capsule, which contains 350 mg AOB-w or the placebo with the same dose. Urine were collected within 48 hours thereafter. The diet was rigorously controlled within 24 hours prior to study till entire study finished. Four mercapturic acid metabolites have been investigated as urinary biomarkers for short-term internal exposure of acrylamide in human

ELIGIBILITY:
Inclusion Criteria:

* Subject has no smoking or drinking hobby

Exclusion Criteria:

* Having any drugs within 7days
* Smoking or drinking
* Pregnant, trying to become pregnant or breast feeding
* Allergic frying foods

Ages: 17 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 110 (Actual)
Dates: Start 2014-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change of four urinary biomarkers of acrylamide | up to 48 hours
  Urine was collected prior to the potato chips meal and 48 hours thereafter, up to 10 urine samples for each participants. Urinary biomarkers of acrylamide were detected by UHPLC-MS/MS.
Change of two hemoglobin adducts of acrylamide | baseline, 3 and 10 days
  Blood samples were collected in 0, 3, 10days after the intake of potato chips meals. Two hemoglobin adducts (AAVal and GAVal) of acrylamide were detected by UHPLC-MS/MS.

SECONDARY OUTCOMES:
Area under the concentration versus time curve (AUC) Of acrylamide urinary biomarkers | baseline, 2, 4, 6, 8, 10, 14, 24, 36 and 48 hours
  Dynamic changes of biomarkers during the specified intervention period, following 10 urine samples in 48 hours thereafter.
Maximum Concentration (Cmax) of Acrylamide Urinary Biomarkers | 48 hours
  Maximum concentration of urinary biomarkers during the specified period, measured by curve fitting tools of Matlab Software.
Time to Peak Concentration (tmax) of Acrylamide Urinary Biomarkers | 48 hours
  Time to Peak Concentration (tmax) of Acrylamide Urinary Biomarkers during the specified period, measured by curve fitting tools of Matlab Software.

IPD SHARING:
Plan to Share IPD: No